CLINICAL TRIAL: NCT00396851
Title: Double Blind Randomized Trial to Compare Gurmar (Gymnema Sylvestre) With Metformin in Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: Indian Council of Medical Research (Other Government); International Clinical Epidemiology Network (INCLEN) TRUST (Network)
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pharma 6/700
Record Dates: First submitted 2006-11-06; First posted 2006-11-08 (Estimated); Last update posted 2006-11-08 (Estimated); Status verified 2006-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

INTERVENTIONS:
Drug: Gurmar
Drug: Metformin

SUMMARY:
The study plans to compare the glucose-lowering effect of gurmar, a herbal preparation, with metformin in patients with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Newly detected type 2 diabetes
* Fasting plasma glucose >126mg/dl
* HbA1c > 7%

Exclusion Criteria:

* Serious comorbid illnesss
* History of drug abuse
* History of recent weight loss

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Bhasin, MD,DM, Study Chair — Post Graduate Institute of Medical Education and Research, Chandigarh; Anil Bhansali, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- PGIMER, Chandigarh, India

REFERENCES:
- [Derived] Gnesin F, Thuesen ACB, Kahler LKA, Madsbad S, Hemmingsen B. Metformin monotherapy for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Jun 5;6(6):CD012906. doi: 10.1002/14651858.CD012906.pub2. PMID 32501595